CLINICAL TRIAL: NCT03537820
Title: Relationship Between Noise Level and Patients Satisfaction in Post Anesthesia Care Units
Brief Title: Noise Impact in the Post-anesthesia Care Unit
Acronym: Post op NOISE
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18016
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: All Surgery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- before nurses formation/installation of a noise warning device: ambulatory or hospitalized patients, who go in post-anesthesia care unit, before nurses formation and installation of a noise warning device
  Interventions: Other: questionnaire
- after nurses formation/installation of a noise warning device: ambulatory or hospitalized patients, who go in post-anesthesia care unit, after nurses formation and installation of a noise warning device
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — questionnaire EVAN-G

SUMMARY:
World health organization recommends noise level should be less than 30db in hospital. However many analysis conclude to an average of 67dB in the post anesthesia care unit. No many studies were reported about noise impact in a post-anesthesia care unit. Only one was published by B.Allaouchiche in 2002. However, noise is a complaint reported by patients and it could be responsible for physiological and psychological troubles. In this prospective study, the main objective is to determine patients' satisfaction in the post anesthesia care unit, before and after installation of a noise warning device. Between the two parts, a short training about noise consequences on health will be presented to nurses. Improvement off anti-noise actions on patient's satisfaction will analysed.

DETAILED DESCRIPTION:
Although the post- anesthesia care unit can be noisy, the effect of noise on patients recovering from anesthesia is unknown. Indeed, many studies are achieved in reanimation or ICU. That's why this prospective study is about patients' satisfaction after their stay in the post-anesthesia care unit. In a first part, noise is just measured with a sound level meter and patients are asked about their experience. Before the second part, during few days, nurses will be informed about noise consequences on heath. With some precaution, a decrease of the sound level in a room (ex: decrease scope alarms, speaking quietly, not slamming the drawer, noise warning device…) will be expected. The main objective is to determine the patient's satisfaction in the post-anesthesia care unit before and after installation of a noise warning device.

ELIGIBILITY:
inclusion criteria :

* patient who have a scheduled surgery in University hospital of Reims
* patient who stay in the post-anesthesia care unit
* patient consenting to participate to the study
* patient older than 18 years

exclusion criteria :

* Emergency surgery
* Patients who have been hearing disorders (notice in the preoperative consultation)
* Patients who have cognitive disorders (notice in the preoperative consultation)
* Patients who have a medical history of ear/cerebral surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with scheduled surgery
Sampling Method: Non-Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
patient's unpleasantness due to the noise | day 1
  visual analog scale EVAN-G

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided